CLINICAL TRIAL: NCT00686738
Title: Validity Verification of Indices Utilizing TGF-b1, NF-kB, PET/CT, and MRS Predicting Response to Neoadjuvant Chemotherapy in Osteosarcoma Patients
Brief Title: Development of Indices Predicting Response to Pre-operative Chemotherapy in Osteosarcoma Patients
Status: Completed | Type: Observational
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Byung-Kiu Park, Head of Center for Pediatric Oncology, National Cancer Center, Korea
Other Study IDs: NCCCTS-07-256
Record Dates: First submitted 2008-05-27; First posted 2008-05-30 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-03

CONDITIONS: Osteosarcoma
Keywords: osteosarcoma; transforming growth factor-beta 1; nuclear factor-kappa B; positron emission tomography/computed tomography; magnetic resonance spectroscopy; predicting response to neoadjuvant chemotherapy
MeSH Terms: conditions — Osteosarcoma; Camurati-Engelmann Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — NF-kB expression status will be determined on initial biopsy and surgically removed tumor specimen.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- A: Study group will be made up of patients hospitalized to National Cancer Center, Korea, aged between 5 and 40 years, and diagnosed with high grade osteosarcoma by histological exam.
  In this group, TGF-b1 measurement, PET/CT and MRS examination at diagnosis, after 1st cycle chemotherapy, and 2nd or 3rd chemotherapy (just before surgery) will be made.
  In addition, evaluation of NF-kB expression status in tumor specimens at diagnostic biopsy and tumor removing surgery will be done.
  The results of above studies will be correlated with the necrosis fractions of the tumor tissues removed by surgery.

SUMMARY:
The purpose of this study is to develop indices predicting response to pre-operative chemotherapy in osteosarcoma patients. Histologic response to pre-operative chemotherapy is very important for the ultimate outcome of osteosarcoma patients. Conventional methods such as CT or MRI evaluating tumor response to chemotherapy is not so efficient in tumors like osteosarcoma. Instead, the investigators will test whether blood TGF-b1 levels, PET/CT findings, MRS findings as well as the level of NF-kB expression in tumor tissues can predict chemotherapy response in osteosarcoma.

DETAILED DESCRIPTION:
We will conduct a prospective trial to verify the validity of indices utilizing TGF-b1, NF-kB, PET/CT, and MRS for predicting response to neoadjuvant chemotherapy in osteosarcoma patients. We assume that changes in plasma TGF-b1 levels, PET/CT and magnetic resonance spectroscopy (MRS) findings during the period of neoadjuvant chemotherapy as well as the initial nuclear NF-kB expression status of tumor biopsy specimen either alone or in combination may predict a chemotherapeutic response determined by histopathologic necrosis fractions of tumors removed. To test this, we will obtain TGF-b1 levels, PET/CT and MRS findings at diagnosis and at follow-up (after first and second/third chemotherapy cycle). Tumor will then be removed. Chemotherapy regimen comprised of various combination of cisplatin, adriamycin, and high-dose methotrexate, ifosfamide, and etoposide. Indices derived from TGF-b1, PET/CT, MRS predicting greater than 90% necrosis fractions will be sought utilizing statistical methods.

ELIGIBILITY:
Inclusion Criteria:

* Karnofsky (over 15 years) or Lansky (less than 15 years) score equal or greater than 50
* Adequate organ functions:

  * GFR>60ml/min/1.73m2
  * EF>50% or SF>28% on echocardiogram
  * ANC>1.5 x 10^9/L
  * platelet>100 x 10^9/L
* Obtainment of informed consents from parents/legal guardians and/or patients

Exclusion Criteria:

* Pregnant or lactating women
* Cardiovascular dysfunction
* History of previous chemotherapy

Ages: 5 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: osteosarcoma patients hospitalized to National Cancer Center, Korea
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2007-02; Primary Completion 2012-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
histopathologic necrosis fractions of surgically removed tumor specimen | 12-17 weeks after starting chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Byung-Kiu Park, M.D., Ph.D., Principal Investigator — Pediatric Oncology Branch, National Cancer Center, Korea
Locations (1):
- National Cancer Center, Goyang-si, Gyeonggi-do, South Korea